CLINICAL TRIAL: NCT07162922
Title: Impact of Intra-abdominal Pressure on Optic Nerve Sheath Diameter During Laparoscopic Cholecystectomy: A Randomized Prospective Study
Brief Title: Optic Nerve Sheath Diameter Changes in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Engin Çetin (Other Government)
Responsible Party: Sponsor-Investigator, Engin Çetin, principal investigator, Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KSH-ANREA-EC-02
Record Dates: First submitted 2025-08-20; First posted 2025-09-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Increased Intracranial Pressure Disorders; Perioperative Complication; Pneumoperitoneum
Keywords: optic nerve sheath,; ultrasonography,; cholesistectomy,; pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 mmHg pressure group (Active Comparator): Patients in this group will undergo laparoscopic cholecystectomy with pneumoperitoneum maintained at 8 mmHg.
  Interventions: Other: 8 mmHg pressure group
- 14 mmHg pressure group (Active Comparator): Patients in this group will undergo laparoscopic cholecystectomy with pneumoperitoneum maintained at 14 mmHg.
  Interventions: Other: 14 mmHg pressure group

INTERVENTIONS:
Other: 8 mmHg pressure group — Laparoscopic cholecystectomy will be performed with intra-abdominal pressure maintained at 8 mmHg during insufflation. Standard anesthesia and surgical protocols will be followed.
  Arms: 8 mmHg pressure group
Other: 14 mmHg pressure group — Laparoscopic cholecystectomy will be performed with intra-abdominal pressure maintained at 14 mmHg during insufflation. Standard anesthesia and surgical protocols will be followed.
  Arms: 14 mmHg pressure group

SUMMARY:
Purpose The goal of this clinical trial is to learn how different intra-abdominal pressures during laparoscopic cholecystectomy affect the optic nerve sheath diameter (ONSD), which is a non-invasive marker of intracranial pressure. The study will also evaluate whether these changes are related to symptoms such as headache, confusion, and nausea after surgery.

Study Design

This is a prospective, randomized, double-blind clinical trial. Patients undergoing elective laparoscopic cholecystectomy will be assigned to one of two groups:

Group 1: pneumoperitoneum at 8 mmHg Group 2: pneumoperitoneum at 14 mmHg ONSD will be measured at several time points before, during, and after surgery using transorbital ultrasonography.

DETAILED DESCRIPTION:
Purpose The aim of this clinical trial is to investigate how different intra-abdominal pressures applied during laparoscopic cholecystectomy affect the optic nerve sheath diameter (ONSD), which serves as a reliable, non-invasive marker of intracranial pressure. The study also seeks to determine whether perioperative ONSD changes are associated with postoperative symptoms such as headache, nausea, and disorientation, as well as with recovery parameters and hemodynamic stability.

Study Design

This is a prospective, randomized, double-blind, interventional clinical trial. Eligible patients scheduled for elective laparoscopic cholecystectomy will be randomized into two groups based on pneumoperitoneum pressure:

Group 1 (Low-pressure group): pneumoperitoneum maintained at 8 mmHg Group 2 (High-pressure group): pneumoperitoneum maintained at 14 mmHg

ONSD will be measured via transorbital ultrasonography at standardized perioperative time points:

T0: Before induction of anesthesia

T1: 30 minutes after initiation of pneumoperitoneum

T2: 5 minutes after extubation

T3: 1 hour postoperatively

T4: 2 hours postoperatively

All ultrasonographic assessments will be performed by a trained investigator blinded to the patient's group allocation.

Participation Patients will receive anesthesia and undergo laparoscopic cholecystectomy according to standard surgical protocols.

Each participant will be randomly assigned to one of the two pneumoperitoneum pressure groups (8 mmHg or 14 mmHg).

After surgery, patients will be observed in the recovery unit. Postoperative symptoms including headache, nausea and vomiting will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* ASA physical status I-II
* BMI < 30 kg/m²
* Scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* Known neurological diseases
* Ocular pathology
* History of elevated intracranial pressure (ICP)
* Pregnancy
* Need for emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-12-21 (Actual); Study Completion 2025-12-21 (Actual)

PRIMARY OUTCOMES:
Effects of Pneumoperitoneum Pressure on ONSD Over Time | T0: Before intubation T1: 30 minutes after the initiation of pneumoperitoneum T2: 5 minutes after extubation T3: 1 hour after extubation T4: 2 hours after extubation
  To compare the effect of two different pneumoperitoneum pressures (8 mmHg vs. 14 mmHg) on optic nerve sheath diameter (ONSD) during laparoscopic cholecystectomy. ONSD will be assessed by measuring changes with transorbital ultrasonography at multiple perioperative time points

SECONDARY OUTCOMES:
Number of participants with postoperative nausea assessed by a standardized 4-point nausea scale | One hour after surgery
  Postoperative nausea will be assessed one hour after surgery using a standardized 4-point scale (0 = no nausea, 1 = mild, 2 = moderate, 3 = severe). The number and proportion of participants with any nausea (score ≥1) will be recorded. Higher scores indicate worse symptoms.
Number of participants with postoperative vomiting within one hour after surgery | One hour after surgery
  Occurrence of vomiting will be recorded during the first postoperative hour. The number and percentage of participants experiencing at least one vomiting episode will be documented (yes/no outcome)
Severity of postoperative headache assessed by Numerical Rating Scale (NRS, 0-10) | One hour after surgery
  Postoperative headache will be evaluated one hour after surgery using a Numerical Rating Scale (NRS), where 0 = no pain and 10 = worst possible pain. Mean NRS scores and the proportion of participants with moderate-to-severe headache (NRS ≥4) will be reported. Higher scores indicate more severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blecha S, Harth M, Schlachetzki F, Zeman F, Blecha C, Flora P, Burger M, Denzinger S, Graf BM, Helbig H, Pawlik MT. Changes in intraocular pressure and optic nerve sheath diameter in patients undergoing robotic-assisted laparoscopic prostatectomy in steep 45 degrees Trendelenburg position. BMC Anesthesiol. 2017 Mar 11;17(1):40. doi: 10.1186/s12871-017-0333-3. PMID 28284189